CLINICAL TRIAL: NCT05905003
Title: Accelerating Medicines Partnership® Schizophrenia Observational Study: Psychosis Risk Evaluation, Data Integration, and Computational Technologies -Data Processing, Analysis, and Coordination Center and Coordination Center
Brief Title: AMP SCZ® Observational Study: PREDICT-DPACC
Acronym: AMP SCZ
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Orygen (Other); Yale University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martha E Shenton, Senior Scientist, Brigham and Women's Hospital
Other Study IDs: 2020P002267; U24MH124629 (NIH); U01MH124631 (NIH); U01MH124639 (NIH)
Record Dates: First submitted 2023-05-17; First posted 2023-06-15 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Clinical High Risk; Psychosis; Remission; Conversion
Keywords: biomarkers; phenotype
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, leukocytes, plasma, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CHR: Clinical High Risk (CHR) for psychosis subjects meeting diagnostic criteria for CHR on the Positive SYmptoms and Diagnostic Criteria for the CAARMS Harmonized with the SIPS (PSYCHS).
- HC: Healthy Control (HC) Subjects

SUMMARY:
The Accelerating Medicines Partnership® Schizophrenia (AMP® SCZ) is a large international collaboration to develop algorithms using a set of clinical and cognitive assessments, multi-modal biomarkers, and clinical endpoints that can be used to predict the trajectories and outcomes of individuals at clinical high risk (CHR) for psychosis and to advance the testing of pharmacological interventions for CHR individuals in need. The goal is to accurately predict which individuals are likely to remit, experience an acute psychotic episode, or have intermediate outcomes that feature persistent attenuated psychotic and/or mood symptoms along with functional impairment. The prediction algorithms will have the potential to serve as early indicators of treatment efficacy in CHR persons.

The AMP SCZ research program is made up of the Psychosis Risk Evaluation, Data Integration, and Computational Technologies - Data Processing, Analysis and Coordination Center (PREDICT-DPACC) and two clinical research networks, the Psychosis-Risk Outcomes Network (ProNET) and the Trajectories and Predictors in the Clinical High Risk for Psychosis Population: Prediction Scientific Global Consortium (PRESCIENT) networks. The two clinical research networks will recruit a large cohort of CHR young people aged 12-30 years (n=1,977) and healthy control (HC) participants (n=640) across 42 participating investigative sites from 13 countries. CHR participants will complete screening, baseline assessments and a battery of follow-up assessments across 18 - 24 months. HC participants will complete screening and baseline assessments and a subset (5 per site) will complete month 2, 12 and 24 visits.

DETAILED DESCRIPTION:
The Accelerating Medicines Partnership (AMP®) is a public-private partnership between the National Institutes of Health (NIH), the U.S. Food and Drug Administration (FDA), the European Medicines Agency, and multiple public and private organizations. The goal of the AMP Schizophrenia (AMP SCZ) program, a multi-continent consortium, is to develop a deep biomarker-informed functional characterization and longitudinal clinical profiling of study participants at clinical high risk (CHR) for psychosis. The data will support the development of algorithms of clinical and biological measures to predict the trajectories and outcomes of CHR individuals to identify enriched CHR patient populations to enable proof of principle intervention studies for early intervention in schizophrenia. These tools will allow the assessment of biomarkers and outcome measures as early indicators of pharmacologic treatment efficacy. See the AMP SCZ website link for a detailed description of study goals (https://www.ampscz.org/about/goals/).

The Accelerating Medicines Partnership® Schizophrenia Observational Study: Psychosis Risk Evaluation, Data Integration, and Computational Technologies Data Processing, Analysis and Coordination Center (AMP SCZ® Observational Study: PREDICT-DPACC) based out of Brigham and Women's Hospital (BWH) and Mass General Brigham (MGB) is one of three research projects supported by the AMP SCZ program.

The AMP SCZ Observational Study: PREDICT-DPACC works with two Clinical High Risk (CHR) research networks (described below) to meet the following goals:

* Capture data from the research networks in a uniform manner.
* Build flexible infrastructure to accommodate multiple data types.
* Develop and refine pipelines that provide rapid data processing (in close to real-time) and quality assurance (QA) and quality control (QC).
* Provide data coordination, management, and monitoring of data.
* Develop powerful and robust stratification tools to identify & validate biomarkers and predict individual outcome trajectories.
* Assist in archiving data and making it publicly available in the NIMH Data Archive (NDA). Please see (https://nda.nih.gov/ampscz/).
* Disseminate information, including tools developed, to the general research community, and provide outreach to the community via a website.

MGB institutions do not provide or enroll participants for this study but serve as the AMP SCZ DPACC for two CHR Research Networks (RNs) where consent and all clinical testing and data collection occur. MGB is a data recipient only, not a data provider. The Mass General Brigham IRB is the IRB of record for the AMP SCZ® Observational Study: PREDICT-DPACC and the IRB status is exempt.

The two CHR research networks (RNs) that also make up the AMP SCZ program are:

The Psychosis-Risk Outcomes Network (ProNET) is based out of Yale University, which serves as the hub for this network and consists of a network of sites in the US, Canada, Europe, and Asia. Northwell Health is the IRB of record for all US sites in the ProNET RN. All foreign ProNET sites submit to their local IRBs.

The Trajectories and Predictors in the Clinical High Risk for Psychosis Population: Prediction Scientific Global Consortium (PRESCIENT), is based out of the Center for Youth Mental Health at the University of Melbourne and at Orygen, Melbourne, Australia, which serves as the hub for this network, and consists of a network of sites in Australia, Europe, and Asia. The Melbourne Health Research Governance and Ethics Office for Research is the IRB of record for all Australian sites in the PRESCIENT research network. European and Asian sites submit to their local IRBs.

Acquisition Sites collect the data and transfer it directly to Brigham and Women's Hospital, which is the main site for the Data Processing Analysis and Coordination Center (DPACC).

See the AMP SCZ website for a searchable map with contact information for all study sites (https://www.ampscz.org/about/map/). Please also see the AMP SCZ website for additional information about the ProNET and PRESCIENT research networks and the PREDICT-DPACC coordination center (https://www.ampscz.org/about/networks-coordination/).

This is a non-interventional study examining clinical trajectories and predictors of outcomes in the CHR population. The CHR cohort and HCs will be assessed with a core set of measures at baseline and 2 months post-baseline, with additional assessments completed at other time points. CHR subjects will be assessed longitudinally for 2 years. Participants who develop first-episode psychosis ('converted' cases) during their study participation will continue to be assessed as scheduled. Measures include clinical, cognitive, neurophysiology, neuroimaging, genetics and fluid biomarkers, speech and facial expression (audio/video recordings are optional), and outcome assessments. Digital assessments such as daily ecological momentary assessment (daily digital diary entries) and passive sensing measurements (actigraphy and geolocation) are optional. See the AMP SCZ website for detailed descriptions of the study design (https://www.ampscz.org/scientists/design/) and protocol (https://www.ampscz.org/wp-content/uploads/2023/01/AMP-SCZ-Protocol-Summary-for-Distribution_24JAN2023.pdf).

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 12 and 30 years old;
* Understand and sign an informed consent (or assent for minors) document;
* Meet diagnostic criteria for CHR from the Positive SYmptoms and Diagnostic Criteria for the CAARMS Harmonized with the SIPS (PSYCHS).

Exclusion Criteria:

* Antipsychotic medication exposure equivalent to a total lifetime haloperidol dose of >50 mg or current antipsychotic medication at time of screening assessment;
* Documented history of intellectual disability;
* Past or current clinically relevant central nervous system disorder;
* Traumatic brain injury that is rated as 7 or above on the Traumatic Brain Injury screening instrument;
* Current or past treated or untreated psychotic episode, as determined using the PSYCHS.

See also the AMP SCZ website link for a description of eligibility criteria (https://www.ampscz.org/participate/eligible/).

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects are recruited and tested at 42 Clinical High Risk research/clinical treatment sites throughout the US, Canada, Australia, Europe, South America, and Asia. The individual sites are part of 2 Research Networks, the Psychosis-Risk Outcomes Network (ProNET) based out of Yale University, and the Trajectories and Predictors in the CHR for Psychosis Population: Prediction Scientific Global Consortium (PRESCIENT) based out of the University of Melbourne/Orygen.
Sampling Method: Non-Probability Sample
Enrollment: 2617 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Conversion to Psychosis | By 24 month follow-up.
  Conversion to psychosis as defined by psychosis threshold criteria on the PSYCHS.

SECONDARY OUTCOMES:
Remission | By 24 month follow-up.
  Recovery from CHR as defined by PSYCHS criteria.
Non-conversion/Non-remission | By 24 month follow-up.
  Continued CHR condition as defined by PSYCHS criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Martha E Shenton, Ph.D., Principal Investigator — Brigham and Women's Hospital/Harvard Medical School; Scott Woods, M.D., Principal Investigator — Yale University; Barnaby Nelson, Ph.D., Principal Investigator — Center for Youth Mental Health at the University of Melbourne/Orygen
Locations (42):
- United States (17):
  - University of California Irvine, Irvine, California
  - University of California Los Angeles, Los Angeles, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Hartford Healthcare, Hartford, Connecticut
  - Yale University/Connecticut Mental Health Center, New Haven, Connecticut
  - University of Georgia, Athens, Georgia
  - Northwestern University, Evanston, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Northwell Health, Queens, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Oregon, Eugene, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Australia (7):
  - HEP and co-located Headspace Adelaide, Adelaide, South Australia
  - Headspace, Craigieburn, Craigieburn, Victoria
  - Headspace, Glenroy, Glenroy, Victoria
  - Headspace Melton, Melton South, Victoria
  - Orygen Specialist Programs, Melbourne, Parkville, Victoria
  - Headspace, Sunshine, Sunshine, Victoria
  - Headspace, Werribee, Werribee, Victoria
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - McGill University, Montreal, Quebec
- Hospital Clínico Universidad de Chile (HCUCH), Santiago, Santiago Metropolitan, Chile
- Shanghai Jiao Tong University, Shanghai, China
- Copenhagen Research Center for Mental Health (CORE), Copenhagen, Denmark
- Germany (3):
  - Klinik für Psychiatrie und Psychotherapie, University of Cologne, Cologne, Brescia
  - The University Hospital Jena, Department of Psychiatry, Jena, Thuringia
  - Ludwig-Maximilians-Universität Munich, Munich
- The University of Hong Kong, Department of Psychiatry, Hong Kong, Hong Kong
- University of Pavia, Pavia, Pavia, Italy
- Early Psychosis Intervention Programme (EPIP) Clinic, Institute of Mental Health, Singapore, Singapore
- South Korea (2):
  - Department of Psychiatry, Chonnam National University Hospital & Mindlink, Gwangju
  - Seoul National University College of Medicine, Seoul
- Instituto de Psiquiatría y Salud Mental Hospital General Universitario Gregorio Marañón, Madrid, Spain
- Treatment and Early Intervention in Psychosis Program (TIPP) & Center for Psychiatric Neuroscience (CNP), Department of Psychiatry, Lausanne University Hospital, Lausanne, Switzerland
- United Kingdom (3):
  - Forward Thinking Birmingham, Birmingham
  - University of Cambridge, Cambridge
  - King's College London, London

IPD SHARING:
Plan to Share IPD: Yes
AMP SCZ will be collecting a wide range of data types as described below:
  * Ascertainment & outcome measures - will be stored as tabular data (multiple formats possible, csv)
  * Neurocognitive measures - will be stored as tabular data (multiple formats possible, csv)
  * EEG data
  * MRI data
  * Audio/Video data
  * Digital Biomarkers (EMA) including
    * Phone Surveys
    * Phone GPS
    * Phone Accelerometry
    * Phone Audio diary
    * Watch/sensor actigraphy (captured by an Axivity device)
  * Genetics & Fluid Biomarkers metadata forms
  Data will include QCed raw data as well as processed data and derivatives. Sensitive data will be identified and separated from non-sensitive data.
  Data sharing will be consistent with subject consent data use limitations.
Supporting Information: Study Protocol
Time Frame: NIMH Data Archive (NDA) Curated Release Environment. Curated releases will be made available to the larger research community approximately every 6 months. The Psychosis Risk Evaluation, Data Integration, and Computational Technologies (PREDICT) Data Processing, Analysis and Coordination Center (PREDICT-DPACC) will be responsible for packaging the data from the project that will be shared in curated releases and submitted to the NDA. This will follow standard NDA procedures with all NDA dictionaries and NDA QA/QC protocols. Data will include QCed raw data as well as processed data and derivatives. Sensitive data will be identified and separated from non-sensitive data. Qualified researchers will need to submit a Data Access Request to the NDA to see these data. The PREDICT-DPACC will not be responsible for granting access to these data on the NDA. NDA may decide to require separate agreements for sensitive vs non-sensitive data.
Access Criteria: For accessing data on the NDA please see https://nda.nih.gov/ampscz/access-data-info.html
URL: https://nda.nih.gov/ampscz/

REFERENCES:
- See also: The website conveys an overview of the aims and activities of the program for consumption by researchers, potential help seeking patients and their families as well as clinicians and clinics looking to update best practice guidelines. — http://ampscz.org
- Available data/document: Individual Participant Data Set — https://nda.nih.gov/ampscz/

DOCUMENTS (4):
  • Study Protocol: ProNET Study Protocol (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT05905003/Prot_000.pdf
  • Study Protocol: PRESCIENT Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT05905003/Prot_001.pdf
  • Informed Consent Form: ProNET CHR ICF (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT05905003/ICF_002.pdf
  • Informed Consent Form: PRESCIENT CHR Self (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT05905003/ICF_003.pdf